CLINICAL TRIAL: NCT06242639
Title: Clinical Acceptability of Metal-ceramic Fixed Partial Dentures Fabricated With Laser Sintering Technique: An up to 7- Year Retrospective Clinical Study
Brief Title: Metal-ceramic Fixed Partial Dentures Fabricated With Laser Sintering
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Selin Çelik Öge, lecturer, Cukurova University
Other Study IDs: Selin Çelik Öge
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Survival, Prosthesis; Clinical Acceptability, Prosthesis
Keywords: metal-ceramic restorations; laser sintering
MeSH Terms: conditions — Prosthesis Failure | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metal-ceramic FPD
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination — clinic and radiographic evaluation

SUMMARY:
The aim of this retrospective clinical study was to evaluate the clinical acceptability of metal-ceramic fixed partial dentures (FPD) manufactured utilizing direct metal laser-sintering technology, taking into account the short-term, medium-term, and long-term outcomes. The Federation Dentaire International (FDI) World Dental Federation criteria were used to evaluate the esthetic, functional, and biological clinical acceptability of the patients who met the inclusion criteria

DETAILED DESCRIPTION:
Objectives: To evaluate the clinical success of laser sintered metal-ceramic restorations throughout several time periods, including the short, medium, and long term.

Materials and methods: Participants who had 3-unit metal-ceramic fixed partial dentures fabricated by laser sintering in the mandibular posterior region between 2014 and 2021 were evaluated. The FDI criteria were used to evaluate the esthetic, functional, and biological clinical acceptability of the patients who met the inclusion criteria. The surface luster was assessed and given a score in the field of esthetic properties. The functional parameters were assessed and rated based on fracture, marginal adaptation, radiographic examination, contact point/food impaction, and patient satisfaction. The biological parameters assessed and rated included tooth vitality, periodontal response, mucosa, and oral health. Following the examinations, each parameter was assigned a score ranging from 1 to 5. (1=Clinically excellent/very good, 2=Clinically good, 3=Clinically satisfactory, 4=Clinically unsatisfactory, 5=Clinically poor) Scoring between 1 and 3 was deemed clinically acceptable, whereas scoring 4 or 5 was deemed clinically unacceptable.

Descriptive statistical analysis was performed for all data.

ELIGIBILITY:
Inclusion Criteria:

* Patients who treated between 2014 and 2021 by prosthodontists at Cukurova University Faculty of Dentistry, Department of Prosthodontics.
* Patients who treated three-unit metal-ceramic fixed partial dentures due to mandibular posterior single tooth deficiency

Exclusion Criteria:

* Patients with any non-vital abutment teeth
* Patients who have severe generalize periodontitis

Ages: 29 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Includes all patients treated by Cukurova University Faculty of Dentistry, Department of Prosthodontics, with laser sintered three-unit metal-ceramic FPD for mandibular posterior single tooth deficiency between 2014 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Surface luster | 1, 3, 5, and 7 years
  The surface luster was scored after visual assessment and short air drying. Score 1 is "Surface luster and surface texture comparable to dental hard tissue/adjacent teeth after air drying" . Score 2 is "Slightly dull surface luster and/or surface texture with minor deviations, e.g., isolated/small marks, pores, and/or voids detectable compared to dental hard tissue/adjacent teeth after air drying" . A score of 3 indicates a dull surface with noticeable deviations such as markings, pores, and voids compared to dental hard tissue/adjacent teeth, even without air drying. Repair is possible". Score 4 is "Localized, displeasing dull surface luster and/or rough surface texture with substantial deviations/multiple pores/voids detectable compared to dental hard tissue/adjacent teeth which can be repaired" . Score 5 indicates a dull or rough surface with significant deviations from dental hard tissue and adjacent teeth. Repair not feasible/reasonable".
Fracture | 1, 3, 5, and 7 years
  Visually and after short air drying, material fracture and retention were rated. Score 1 represents complete restoration without deficiencies after air drying. No cracks, chipping/delamination, or bulk material breakage". Score 2 says, "Restoration is completely present with minor deficiencies detectable after air drying, e.g., insignificant material chipping or one hairline crack" . Score 3 indicates restoration with visible defects, such as hairline fractures or material loss (chipping), even without air drying. Material loss can be addressed by refurbishing if necessary. Score 4 indicates serious fracture and retention issues, such as chipping/delamination, bulk fracture, or partially loose/lost repair. Repair is feasible. Lost indirect restoration, which can be reconstructed, is examined. Scoring 5 indicates serious deficiencies, such as widespread delamination, many bulk fractures, or mostly lost repair. No repair possible/reasonable".
Marginal adaptation | 1, 3, 5, and 7 years
  Marginal gaps are assessed by visual examination, short air drying, and 250 µm probes. Score 1 indicates "Optimal marginal adaptation of the restoration to tooth hard tissue following air drying. No little gap detected by gentle probing". Score 2 indicates small adaption deficiencies after air drying. A little, superficial gap or ditching. 3 indicates, "Distinct deficiencies of marginal adaptation without air drying: marginal gap(s) or ditching (width <250 µm and/or depth <2 mm)" . Score 4 indicates serious marginal adaption deficiencies: width ≥250 µm and/or depth ≥2 mm margin gaps. Partially lost restoration. Repair is feasible". Score 5 indicates substantial marginal adaption impairment: width ≥250 µm and/or depth ≥2 mm. Complete loose/lost restoration. No repair possible/reasonable".
Radiographic evaluation | 1, 3, 5, and 7 years
  Restorations with no pathology on radiographs were considered score 1. Restorations with secondary caries, apical pathology, fracture, and tooth/restoration loss were recorded as score 5.
Contact point/Food impaction | 1, 3, 5, and 7 years
  Proximal contact point was carried out by using visual examination and 25-50-100 µm blades. Score 1 means, "Ideal contact point: 25-µm metal blade can pass through proximal contact". Score 2 means, "Slightly weak contact point: 50-µm metal blade can pass through proximal contact". Score 3 means, "Oversized contact point or excessive material: 25-µm metal blade cannot pass through proximal contact". Score 4 means, "Severely weak contact point: 100-µm metal blade can pass through proximal contact or unintended interlocked contact point". Score 5 means, "Severely weak contact point: 100-µm metal blade can easily pass through proximal contact or unintended interlocked contact point (impossible to pass)".
Patient's view | 1, 3, 5, and 7 years
  Patient comments were attentively listened to and recorded. Score 1 means, "Entirely satisfied with esthetics and function". Score 2 means, "Satisfied". Score 3 means, "Minor criticism but no adverse clinical effects". Score 4 means, "Desire for improvement". Score 5 means, "Completely dissatisfied and/or adverse effects".
Tooth vitality | 1, 3, 5, and 7 years
  The teeth were assessed for loss of vitality and assigned scores. Score 1 means, "Normal vitality". Score 5 means, "Intense, acute pulpitis or non vital tooth. Endodontic treatment is necessary and restoration has to be replaced".
Periodontal response | 1, 3, 5, and 7 years
  The presence of plaque, acceptable/unacceptable plaque level and accompanying inflammation, pocket formation, gingival bleeding on probing, and severe acute/chronic periodontitis were all examined to determine the periodontal response and compared to a reference tooth. Score 1 means, "No plaque, no inflammation, no pockets". Score 5 means, " Severe / acute gingivitis or periodontitis".
Adjacent mucosa | 1, 3, 5, and 7 years
  Visual examination was used to assess the condition of the mucosa around the restoration. Score 1 means, "Healthy mucosa adjacent to restoration". Score 5 means, "Suspected severe allergic, lichenoid or toxic reaction".
Oral and general health | 1, 3, 5, and 7 years
  The existence of any irritation and allergic, lichenoid, or toxicological reactions, and to determine the degree of these reactions. Score 1 means, "No oral or general symptoms". Score 2 means, "Minor transient symptoms of short duration; local or generalized". Score 3 means, "Transient symptoms, local and/or general". Score 4 means, "Persisting local or general symptoms of oral contact stomatitis or lichen planus or allergic reactions. Intervention necessary but no replacement". Score 5 means, "Acute/severe local and/or general symptoms".

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova Univeristy, Adana, Turkey (Türkiye)